CLINICAL TRIAL: NCT04308382
Title: Evaluation of a Corporate Wellness Program
Status: Completed | Type: Observational
Sponsor: Ohio University (Other)
Collaborators: Memorial Health System (Other)
Responsible Party: Principal Investigator, David Drozek, Associate Professor, Ohio University
Other Study IDs: 20-X-6
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease | interventions — Risk Assessment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Health Risk Assessment — Heath Risk Assessment consists of:
  * Survey to include questions about physical activity, stress, hope, household hunger and demographics.
  * Lipid panel and HbA1c
  * Height and Weight, blood pressure and resting pulse

SUMMARY:
The purpose of this project is to determine the effectiveness of the corporate wellness program at Memorial Health System (MHS) in regards to:

1. Improvement of health of employees
2. Savings on health care expenses

The corporate wellness program itself is not the object of the study, but rather the results of the program are the focus. The program will be a dynamic process, changing over time to address the needs of the hospital system employees.

This study will look at the effects of the program as a whole to impact employee health and the cost of healthcare. This study will also evaluate individual components of the program (physical activity, stress management, etc) to determine specific benefits of those components to those who participate.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of a corporate wellness program to improve the health of its employees and to save healthcare costs.

Many studies have been done evaluating the effectiveness of corporate wellness programs. Over the past 30 years, multiple iterations of corporate wellness programs have been utilized, causing a continual shift in philosophy and implementation. The current program is following closely the model instituted by Cleveland Clinic, utilizing recommendations and tools provided by the CDC and WELCOA via their web sites and publications.

Description of Program to be Evaluated MHS is initiating a corporate wellness program to be offered to all adult employees. The program will include a health risk assessment (HRA), which is the minimum required for enrollment in the program, as well as many additional optional benefits, such as access to exercise equipment, personal coaches, stress management classes, etc. There will also be corporate wide changes to the environment to include food options in the cafeteria and vending machines.

The HRA will be offered annually, and before and after completion of specific activities offered by the wellness program.

The HRA includes a survey, which requires about 30 minutes to complete, lab evaluation and biomarkers.

Research to Evaluate the Program As people are enrolling in the wellness program on line, participants will be invited to participate in this study. People can participate in the wellness program without participating in this study.

The invitation to participate will provide a brief description of the study and a link which will take them to the consent. Once consented, there will be a link to return to the on line program enrollment. They will have the option to email members of the research team with any questions or to request a paper version of the consent and survey.

They may decline study participation, without any penalty, and will be allowed to participate in the wellness program as would anyone who is participating in the study.

There will be an option to use a paper consent. If a paper consent is utilized, these will be collected by the research team. Paper consents will then be stored in a secure location at MHS.

To participate, subjects will also be asked to sign a study specific HIPAA authorization form allowing access to personal health information to be utilized for the study.

Data collected for this study will be maintained with multilevel encryption; devices and cloud storage will be encrypted. Data will need to be identified to allow collation of data from various sources.

For the evaluation of absenteeism and health claims data, aggregated de-identified data for groups of subjects will be requested from HR. These groups will be determined by level of participation in various wellness activities.

The data will be analyzed by the research team to determine overall effectiveness in improving health and reducing health care expenses, as well as looking for correlations with specific variables (age, gender, participation in particular components of the program, etc.)

It is anticipated that aggregated de-identified results will be presented publicly in the form of abstracts, posters and publication.

ELIGIBILITY:
Inclusion Criteria:

-adult employee of Memorial Health System, or spouse of an employee who is participating in the employee wellness program

Exclusion Criteria: NA

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult employees of the Memorial Health System.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Health Care Expenditures | 20 years
  Cost for health care as a corporation

SECONDARY OUTCOMES:
Body Mass Index of employees | 20 years
  Calculated based on manually measured height (feet and inches) and weight (pounds)
Hemoglobin A1c of employees | 20 years
  measured in %
Blood pressure | 20 years
  measured in mm Hg with a sphygmomanometer while at rest
Total cholesterol | 20 years
  laboratory blood analysis, reported in mg/dl
Low density lipoprotein (LDL) cholesterol | 20 years
  laboratory blood analysis, reported in mg/dl
High density lipoprotein (HDL) cholesterol | 20 years
  laboratory blood analysis, reported in mg/dl
Triglycerides | 20 years
  laboratory blood analysis, reported in mg/dl
Level of physical activity | 20 years
  Are you able to walk a mile without significant pain or discomfort? ❒ Yes ❒ No
  In the past 7 days, how many days did you exercise? ______ days
  On days when you exercised, for how long did you exercise (in minutes)? ❒______ minutes per day
  ❒ Does not apply
  How intense was your typical exercise?
  * Light (like stretching or slow walking)
  * Moderate (like brisk walking)
  * Heavy (like jogging or swimming)
  * Very heavy (like fast running or stair climbing)
  * I am currently not exercising
Hope | 20 years
  Hearth Hope Index
Mood | 20 years
  Patient Health Questionnaire-4 (PHQ-4), higher score is more abnormal
Tobacco use | 20 years
  In the last 30 days, have you used tobacco? ❒ Yes ❒ No Smoked? ❒ Yes ❒ No Used a smokeless tobacco product? ❒ Yes ❒ No
  If Yes to any of the above, would you be interested in quitting tobacco use within the next month?
  ❒ Yes ❒ No
Alcohol use | 20 years
  In the past 7 days, on how many days did you drink alcohol? ______ days
  On days when you drank alcohol, how often did you have:
  * If you are a man: 5 or more alcoholic drinks on one occasion?
  * If you are a woman: 4 or more alcoholic drinks on one occasion?
    * Never
    * Once during the week
    * 2-3 times during the week
    * More than 3 times during the week
    * Doesn't apply to me
  Do you ever drive after drinking, or ride with a driver who has been drinking?
  ❒ Yes ❒ No
Diet composition | 20 years
  Questions concerning food types based on a 7 day dietary recall
Food availability | 20 years
  Household Hunger scale
Readiness to Change | 20 years
  On a scale of 1-10, how ready are you to participate in a lifestyle change (diet change, exercise, stress management, control of tobacco, alcohol, etc.) to help improve your health?
  1 being not ready at all, 10 being extremely ready _________
  On a scale of 1-10, how confident are you that by participating in a lifestyle change program that you will be successful?
  1 being not confident at all, 10 being extremely confident _________
Absenteeism | 20 years
  days absent per year

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
De-identified, aggregated data will be made available.